CLINICAL TRIAL: NCT07318337
Title: Effect of Drospirenone-Ethinyl Estradiol (20µg) in Comparison to Drospirenone-Ethinyl Estradiol (30µg) on Free Androgen Index in Polycystic Ovary Syndrome
Brief Title: Effect of Drospirenone-Ethinyl Estradiol (20microgram vs 30 Microgram) on Free Androgen Index in PCOS
Acronym: PCOS FAI CHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mst.Sumyara Khatun (Other)
Collaborators: Bangladesh Medical University (Other)
Responsible Party: Sponsor-Investigator, Mst.Sumyara Khatun, Medical Officer, Bangladesh Medical University
Organization: Bangladesh Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5162
Record Dates: First submitted 2025-12-23; First posted 2026-01-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: PCOS (Polycystic Ovary Syndrome)
Keywords: PCOS; COC; Free androgen index; Drospirenone Ethinyl Estradiol
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Intervention Model Description: Quasi Experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): participants received 1 tablet Drospirenone-Ethinyl Estradiol(20µg), once daily for 24 days followed by 4 days placebo for 3cycles
  Interventions: Drug: Drospirenone Ethinyl Estradiol (20 microgram)
- Comparator arm (Active Comparator): Comparator arm received Drospirenone-Ethinyl Estradiol (30 µg) once daily for 21 days followed by 7 days placebo for 3 cycles
  Interventions: Drug: Drospirenone Ethinyl Estradiol (30 microgram)

INTERVENTIONS:
Drug: Drospirenone Ethinyl Estradiol (20 microgram) — 1tablet for consecutive 24 days followed by 4 days placebo for 3 months
  Arms: Experimental arm
Drug: Drospirenone Ethinyl Estradiol (30 microgram) — once daily for 21 days followed by 7 days placebo for 3 months
  Arms: Comparator arm

SUMMARY:
Combined hormonal contraceptive (CHC) improves androgen parameter in women with PCOS. High-dose CHC increases insulin resistance, whereas low dose CHC has minimal effects on carbohydrate metabolism. This quasi experimental study was conducted to compare the effects of Drospirenone-Ethinyl Estradiol (20µg) to that with Drospirenone-Ethinyl Estradiol (30µg) on free androgen index (FAI) in polycystic ovary syndrome. Medication was given for 3 months. FAI, HOMA-IR was measured in baseline and after treatment and results were compared.

DETAILED DESCRIPTION:
This quasi-experimental study was conducted in the Department of Reproductive Endocrinology and Infertility, Bangladesh Medical University (BMU), from July 2024 to June 2025. Ethical clearance was obtained from the Institutional Review Board (Approval no. 5162). A total number of 60 subfertile women with PCOS (according to Rotterdam criteria) (Oligomenorrhoea-defined as delayed menses >35 days or <8 spontaneous menstrual cycle/ year, hyperandrogenism (hirsutism using modified Ferriman-Gallway score of >8, polycystic ovarian morphology on ultrasonography >12 follicles in each ovary measuring 2-9 mm in diameter and/or increased ovarian volumes > 10 cm3) and aged from 20 to 35 years were enrolled in the study. Exclusion criteria encompassed: contraindication to CHC (History of thromboembolic disorder, cerebrovascular disease, coronary artery disease, carcinoma of breast or other estrogen dependent neoplasm, undiagnosed abnormal genital bleeding, known or suspected pregnancy, benign or malignant liver neoplasm, cholestatic jaundice on previous pregnancy, abnormal liver and renal function, uncontrolled DM and HTN, dyslipidemia, history of migraine with focal aura), recent use of androgen and anti-androgens within 3 months, BMI ≥30 kg/m2,oligovulation other than PCOS. Sampling was done by convenient sampling.

The patients were explained in details regarding the objectives, rationale and potential benefits of the study and were counseled regarding the drugs and unexpected side-effects. An informed written consent was taken.

Data was collected through interview, physical examinations and laboratory investigations. Baseline clinical, endocrine and biochemical variables were measured.Laboratory investigations like fasting insulin(determined by chemiluminescent microparticleimmunoassay-CMIA)), fasting blood glucose (done by enzymatic method using commercially available reagent kit), total testosterone (Chemiluminescence immunoassay by LIAISON XL Analyzer), SHBG (determined by DiaSorin LIAISON SHBG assay -Chemiluminescence immunoassay) were done.Blood samples were collected in the early morning, after an overnight fasting of 10 hours, for the measurement of fasting insulin and fasting glucose level.

Participants were divided into two groups without randomization by their alternate day of attendance. Interventional groupreceived DRSP-EE (20 µg) 1tablet for consecutive 24 days followed by 4 days placebo whilecomparatorgroup received DRSP-EE (30 µg) once daily for 21 days followed by 7 days placebo for 3 cycles.All participants were instructed not to take any other medications during the study except after consulting the physician. Patients were called every month over telephone to check for compliance or any side effects.

After 3 months of treatment, blood samples were taken for biochemical studies and FAI, HOMA-IR were calculated. Comparison was made between the effect of DRSP-EE (20 µg) and DRSP-EE (30 µg) in subfertile women with polycystic ovary syndrome.

The mean ± SD values were calculated for continuous variables and percentages were calculated for categorical variables.When the data is not normally distributed then Median (IQR) values were calculated for continuous variables,Mann-Whitney U test was used to compare the medians of two independent groups, Wilcoxon signed rank sum test was used for quantitative variables. For comparing categorical data, the Chi-square (x2) test was performed. Comparison of quantitative variables between the study groups was done using unpaired t-test for independent samples when they are normally distributed. Paired t-test was used for quantitative variables within the group, when compared pre-treatment vs post treatment. P values <0.05 was considered as statistically significant.Statistical analyses were carried out by using the Statistical Package for Social Sciences version 26.0 for Windows.

ELIGIBILITY:
Inclusion Criteria: •Age:20-35 years

* Diagnosed case of PCOS patients according to Rotterdam criteria
* women with PCOS

Exclusion Criteria:

* Contraindication of OCP such as history of thromboembolic disorder, cerebrovascular disease, coronary artery disease, carcinoma of breast or other estrogen dependent neoplasm, undiagnosed abnormal genital bleeding, known or suspected pregnancy, benign or malignant liver neoplasm, cholestatic jaundice on previous pregnancy, abnormal liver and renal function, uncontrolled DM and HTN, dyslipidemia, history of migraine with focal aura
* Recent use of androgen and antiandrogens within 3months
* BMI>30kg/m2
* Cause of oligovulation other than PCOS

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Free Androgen Index | 12 weeks
  Free Androgen index was calculated from serum total testosterone and sex hormone binding globulin

SECONDARY OUTCOMES:
HOMA-IR | 12 weeks
  HOMA-IR was calculated from serum fasting glucose and serum fasting insulin

CONTACTS AND LOCATIONS:
Overall Officials: Shakeela Ishrat, FCPS, Study Director — Bangladesh Medical University
Locations (1):
- Bangladesh Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rajashekar S, Giri Ravindran S, Kakarla M, Ausaja Gambo M, Yousri Salama M, Haidar Ismail N, Tavalla P, Uppal P, Mohammed SA, Hamid P. Spironolactone Versus Oral Contraceptive Pills in the Treatment of Adolescent Polycystic Ovarian Syndrome: A Systematic Review. Cureus. 2022 May 25;14(5):e25340. doi: 10.7759/cureus.25340. eCollection 2022 May. PMID 35774693
- [Result] Bhattacharya SM, Jha A, DasMukhopadhyay L. Comparison of two contraceptive pills containing drospirenone and 20 mug or 30 mug ethinyl estradiol for polycystic ovary syndrome. Int J Gynaecol Obstet. 2016 Feb;132(2):210-3. doi: 10.1016/j.ijgo.2015.06.065. Epub 2015 Nov 6. PMID 26613823
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26613823/